CLINICAL TRIAL: NCT01049126
Title: Retrospective Case Study to Determine the Correlation of Patient Outcome to the ChemoFx Assay in Cases With Late Stage Endometrial Cancer
Brief Title: Retrospective Case Study Examining Patient Outcomes Compared to the ChemoFx Assay in Endometrial Cancer Patients
Status: Completed | Type: Observational
Sponsor: Precision Therapeutics (Industry)
Responsible Party: Holly Gallion, MD, Precision Therapeutics
Other Study IDs: PT-106
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Endometrial Cancer
Keywords: Late Stage
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Late stage endometrial cancer
  Interventions: Other: ChemoFx

INTERVENTIONS:
Other: ChemoFx — Chemoresponse Marker Assay

SUMMARY:
The purpose of this study is to assess the relationship of assay sensitive patients versus assay resistant patients with progression free survival.

DETAILED DESCRIPTION:
This is a multicenter, retrospective chart review study of de-identified drug response marker results and a limited data set of clinical outcome data. Data from approximately 70 cases will be collected from approximately 10 study sites and correlated to the ChemoFx drug response marker results. The outcome of progression free survival will be defined as the period of time between the first dose of chemotherapy following the report of the marker result until clinical progression or death. Objective response will be measured from the first dose of chemotherapy following the report of the marker result until progression or change in therapy. Overall Survival will be measured from the start of chemotherapy to the actual date of death.

ELIGIBILITY:
Inclusion Criteria:

* Case has an original pathology report showing stage III, IIIa, IIIb, IIIc, IV, IVa, IVb, or recurrent endometrial cancer.
* Case includes a pathology or cytology report from initial diagnosis showing disease of one or more of the following histologic epithelial cell types: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, transitional cell carcinoma, clear cell carcinoma, or adenocarcinoma, not otherwise specified (N.O.S.).
* Case has been identified for pattern of response evaluation.
* Case must have a commercial ChemoFx drug response marker final report.

Exclusion Criteria:

* Cases of patients who were deceased prior to 1 cycle of chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 70 cases of late stage endometrial cancer that have had ChemoFx drug response marker results from August 2007 to January 31, 2009 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Gallion, MD, Study Chair — Vice President, Clinical Affairs
Locations (1):
- Precision Therapeutics, Inc., Pittsburgh, Pennsylvania, United States